CLINICAL TRIAL: NCT03589534
Title: Home Pregnancy Test Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROTOCOL-0972
Record Dates: First submitted 2018-06-06; First posted 2018-07-18 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-07

CONDITIONS: Pregnancy Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnancy test (Other): pregnancy tests
  Interventions: Diagnostic Test: home pregnancy test

INTERVENTIONS:
Diagnostic Test: home pregnancy test — Each participant will use 4 different home pregnancy tests

SUMMARY:
This study will evaluate consumer preference and consumer results from a number of commercially available home pregnancy tests.

The study is being conducted as a formal assessment home pregnancy tests sold in Western Europe.

DETAILED DESCRIPTION:
The study will be conducted in two parts:

Part 1: Volunteers representative of pregnancy test users will use a range (4 of 7 different tests being evaluated) in their own home to gain usability data. All products will be used according to their instructions for use which, where required, will be translated into English prior to the study start. A study questionnaire will be completed after each test is used.

Part 2: The volunteers will attend the study site soon after completing their last home test and be required to read randomised results of tests conducted by study technicians (pregnant and not pregnant) to gain an understanding of their ability to correctly read results of the tests. The technician will also read and record the test results to enable both the laboratory agreement (technician read) and the consumer readability to be determined and compared for each product.

Each volunteer will be required to provide a urine sample for determining pregnancy status and quantitative urinary hormone measurement (this is done to confirm the result obtained at home using the HPTs).

At the end of the testing period the volunteers will also be asked to rank the four products they have used in the study, based on a series of statements regarding usability and readability of the tests

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-45 years
* Willing to give informed consent
* Willing to conduct a personal home pregnancy test and reveal their pregnancy status

Exclusion Criteria:

* Currently or previously employed by SPD, Alere, Unipath, P&G, Abbott, or affiliates
* Has an immediate relative* currently or previously employed by SPD, Alere, Unipath, P&G, Abbott or affiliates
* Taken a hormonal preparation containing hCG in the last month, e.g. Pregnyl®
* Recently miscarried and yet to have 2 complete menstrual cycles before study start

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
1. Demonstration of volunteer preference for a HPTs. | 1 week
  • The cumulative scores on a 7-point likert scale for ease of use questions on the device usability at home questionnaire, where 1 equals very good and 7 equals very poor for each attribute.
2. Demonstration of volunteer readability of HPTs | 1 week
  • The cumulative scores on a 7-point likert scale for readability questions on the device readability at SPD questionnaire, where 1 equals very easy and 7 equals very difficult for each attribute.
3. Demonstration of consumer preference for a HPT | 1 week
  • The ranking of each Home Pregnancy Test in order of preference

SECONDARY OUTCOMES:
1. Accuracy of reading | 1 week
  The per cent agreement (accuracy) between the result read by the volunteer and true result for each standard tested (i.e 0 hCG will be not pregnant and 25mIU/ml hCG will be pregnant) for each Home pregnancy test evaluated.
Agreement of reading | 1 week
  The agreement between volunteer home pregnancy test results and those of a technician testing the same urine standard (volunteer vs. technician test result)

CONTACTS AND LOCATIONS:
Locations (1):
- SPD Development Company Ltd., Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boxer J, Weddell S, Broomhead D, Hogg C, Johnson S. Home pregnancy tests in the hands of the intended user. J Immunoassay Immunochem. 2019;40(6):642-652. doi: 10.1080/15321819.2019.1671861. Epub 2019 Sep 26. PMID 31556778